CLINICAL TRIAL: NCT06120387
Title: Combined Postoperative Radiotherapy With Kidney Sparing Surgery for Locally Advanced High-risk Ureteral Cancer
Status: Recruiting | Type: Observational
Sponsor: Xuesong Li (Other)
Responsible Party: Sponsor-Investigator, Xuesong Li, Department of Urology, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: LUXUS3.0
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Locally Advanced; Urothelial Carcinoma Ureter
Keywords: upper tract urothelial carcinoma; Radiotherapy; Kidney sparing surgery; Locally advanced; Ambispective cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney sparing surgery+Postoperative radiotheray cohort: Kidney sparing surgery+Postoperative radiotheray cohort
  Interventions: Radiation: Kidney sparing surgery+Postoperative radiotheray
- Radical surgery cohort: Preoperative CT/MRI, chest CT and other examinations are performed to determine the stage of the patient's disease. The surgical plan is the same as the current conventional treatment. After surgery, there is no restriction on the use of postoperative adjuvant chemotherapy or postoperative adjuvant radiotherapy according to the patient's pathological stage and the patient's wish.
  Interventions: Procedure: Radical surgery

INTERVENTIONS:
Procedure: Radical surgery — Radical nephroureterectomy
  Groups: Radical surgery cohort
Radiation: Kidney sparing surgery+Postoperative radiotheray — Kidney sparing surgery+Postoperative radiotheray
  Groups: Kidney sparing surgery+Postoperative radiotheray cohort

SUMMARY:
In this study, we propose to conduct an ambispective study to analyze the safety of preserved renal unit surgery combined with postoperative adjuvant radiotherapy in patients with limited stage ureteral cancer with high risk factors, and the efficacy analysis compared with traditional radical surgery. It is hoped that a treatment method that preserves patients' renal function to improve the tolerance of subsequent drug therapy without decreasing the effect of tumor treatment can be achieved in patients with high-risk factors.

ELIGIBILITY:
Inclusion Criteria:

- 1) Ureteral cancer patients with high-risk factors (high-risk factors define multifocal; G3; T2-4); surgery may be performed with patients undergoing partial terminal ureteral resection or radical nephroureterectomy 2)Age ≥18 years; 3)Completion of abdominopelvic CT 4 weeks before enrollment to exclude distant metastasis and regional lymph node metastasis.

4) Patients did not have other malignant neoplastic diseases in the last 5 years except for non-melanoma of the skin and ductal carcinoma in situ of the breast; Willing to participate in perfecting the necessary examinations and follow-up for the sake of the study, and willing to provide written informed consent.

Exclusion Criteria:

* 1) Distant metastasis or retroperitoneal lymph node metastasis (N+) had been detected at the time of surgery; R2 resection patients; history of bladder cancer; 2) History of pelvic and abdominal radiotherapy; history of inflammatory bowel disease; history of systemic chemotherapy; 3) Pregnant women or breastfeeding women; or women of childbearing potential who are not practicing reliable contraception; (4) The presence of active infections in those with pre-existing or coexisting bleeding disorders 5) clinically significant cardiac disease (e.g., hypertension controlled with medications, unstable angina, New York Heart Association (NYHA) class ≥II congestive heart failure, unstable symptomatic arrhythmias, or class ≥II peripheral vascular disease); 6) Psychological, family, and social factors leading to lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ureteral cancer patients with high-risk factors (high-risk factors define multifocal; G3; T2-4)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2028-11-09 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival (LRFS) | 1-year, 3-year and 5-year
  Local recurrence
Renal Function Indicators | Perioperation and peri-treatment
  eGFR, Crea

SECONDARY OUTCOMES:
Metastasis free survival (MFS) | 1-year, 3-year and 5-year
  Distant metastasis
Overall survival (OS) | 1-year, 3-year and 5-year
  Overall survival
Intravesical and contralateral recurrence free survival(IRFS and CRFS) | 1-year, 3-year and 5-year
  Intravesical and contralateral recurrence free survival
Adverse effects (AE) | Perioperation and peri-treatment
  Adverse effects

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Departmeng of Urology, Peking University First Hospital, Beijing
  - Department of Radiotherapy Oncology, Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roupret M, Seisen T, Birtle AJ, Capoun O, Comperat EM, Dominguez-Escrig JL, Gurses Andersson I, Liedberg F, Mariappan P, Hugh Mostafid A, Pradere B, van Rhijn BWG, Shariat SF, Rai BP, Soria F, Soukup V, Wood RG, Xylinas EN, Masson-Lecomte A, Gontero P. European Association of Urology Guidelines on Upper Urinary Tract Urothelial Carcinoma: 2023 Update. Eur Urol. 2023 Jul;84(1):49-64. doi: 10.1016/j.eururo.2023.03.013. Epub 2023 Mar 24. PMID 36967359
- [Background] Li HZ, Li X, Gao XS, Qi X, Ma MW, Qin S. Oncological Outcomes of Adjuvant Radiotherapy for Partial Ureterectomy in Distal Ureteral Urothelial Carcinoma Patients. Front Oncol. 2021 Sep 30;11:699210. doi: 10.3389/fonc.2021.699210. eCollection 2021. PMID 34660268
- [Background] Arcangeli G, Arcangeli S, Strigari L. A systematic review and meta-analysis of clinical trials of bladder-sparing trimodality treatment for muscle-invasive bladder cancer (MIBC). Crit Rev Oncol Hematol. 2015 Apr;94(1):105-15. doi: 10.1016/j.critrevonc.2014.11.007. Epub 2014 Dec 4. PMID 25541350